CLINICAL TRIAL: NCT04667338
Title: Observational, Multicentre, Cross-sectional Study to Describe Diagnosis and Treatment Patterns in Narcolepsy Patients in Real Life Practice in Spain
Brief Title: A Study to Collect Information of People With Narcolepsy in Spain
Acronym: SOMNUS
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-994-5001; U1111-1259-8720 (Registry Identifier: WHO)
Record Dates: First submitted 2020-12-09; First posted 2020-12-14 (Actual); Results first posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-07

CONDITIONS: Narcolepsy
Keywords: Drug Therapy
MeSH Terms: conditions — Narcolepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Narcolepsy Type 1: Participants with confirmed diagnosis of narcolepsy type 1 (NT1) defined by the International Classification of Sleep Disorders, Third Edition (ICDS-3) will be observed for up to 16 months.
- Narcolepsy Type 2: Participants with confirmed diagnosis of narcolepsy type 2 (NT2) defined by the ICDS-3 will be observed for up to 16 months.

SUMMARY:
This study aims to review information of people with a sleep condition called narcolepsy. Narcolepsy is a condition that causes extreme sleepiness during the day including falling asleep suddenly. Study doctors will review the medical records of the participants from sleep clinics in Spain. They will do this from 1 year before the participant was diagnosed with narcolepsy up to the start of this study.

Participants will visit the sleep clinic once. During this visit, the study doctors will carry out a short medical exam. Participants will also complete a few questionnaires during this visit. If participants cannot visit the clinic for any reason, the clinic staff will arrange a phone call instead.

DETAILED DESCRIPTION:
This is a non-interventional, cross-sectional study with retrospective medical chart review conducted in public and private Spanish sleep clinics, to describe the management of adult participants diagnosed with narcolepsy defined by ICDS-3 in real world practice.

This study will enroll approximately 196 participants (137 with NT1 and 59 with NT2). Participants will be enrolled in 2 cohorts:

* Cohort A: NT1 Participants
* Cohort B: NT2 Participants

The data will be collected retrospectively through clinical records and at study visit (clinical and demographic data, and participant related outcomes [PRO]) in an electronic case report form (eCRF).

This multi-center study will be conducted in Spain. The overall duration of this study is approximately 24 months. Participants will attend a single visit in the participating centers. In the event of a possible outbreak of coronavirus disease 2019 (COVID-19) participants will have a telepathic visits, the invitation to participate, the obtention of participant's informed consent and the collection of participant's questionnaires will be carried out remotely (by phone or via email).

ELIGIBILITY:
Inclusion Criteria:

1. With confirmed diagnosis of narcolepsy defined by ICDS-3.
2. With at least 1-year follow-up with data available at the participating site after initial narcolepsy diagnosis and before study inclusion.
3. With data available at the participant site at least 1-year before first narcolepsy diagnosis.
4. Capable to fulfill the study questionnaires.

Exclusion Criteria:

1. Participating in a clinical trial (less than or equal to [<=] 12 months).
2. With any serious degenerative disease (Alzheimer, Parkinson or epilepsy) or psychiatric condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with confirmed diagnosis of narcolepsy defined by ICDS-3.
Sampling Method: Non-Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2022-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/602118de84b336001e9395c6

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 12 investigative sites in Spain from 18 February 2021 to 04 November 2022.
Pre-assignment Details: This is a non-interventional, retrospective (utilizing existing data from the medical records of patients), cross-sectional study with only one visit, of 214 patient records 210 participants were selected and considered evaluable for this study. 2 participants were not classified as either narcolepsy type 1 (NT1) or narcolepsy type 2 (NT2) and other 2 participants did not fulfil inclusion criteria and were not considered evaluable for this study.
Groups:
- Narcolepsy Type 1: Participants with confirmed diagnosis of NT1 defined by the International Classification of Sleep Disorders, Third Edition (ICDS-3) were observed for up to 16 months.
- Narcolepsy Type 2: Participants with confirmed diagnosis of NT2 defined by the ICDS-3 were observed for up to 16 months.
Period: Overall Study
Arm/Group | Narcolepsy Type 1 | Narcolepsy Type 2
Started | 157 | 53
Naive: Untreated (Participants with narcolepsy who were not treated with any pharmacological treatment from diagnosis to study visit (up to 12 months).) | 8 | 4
Treated (Participants with narcolepsy who were treated with any pharmacological treatment from diagnosis to study visit (up to 12 months).) | 149 | 49
Completed | 157 | 53
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who met the eligibility criteria and participated in the study were included in the study population.
Groups:
- Narcolepsy Type 1: Participants with confirmed diagnosis of NT1 defined by the ICDS-3 were observed for up to 16 months.
- Total: Total of all reporting groups
Arm/Group | Narcolepsy Type 1 | Narcolepsy Type 2 | Total
Number analyzed (Participants) | 157 | 53 | 210
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.2 (13.9) | 42.6 (13.0) | 41.6 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 22 | 101
  Male | 78 | 31 | 109
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 147 | 50 | 197
  Hispanic | 7 | 3 | 10
  Asian / Oriental | 1 | 0 | 1
  Other | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Categorized Based on Treatment by Narcolepsy Type Since Diagnosis up to Study Visit
Description: Percentage of participants with narcolepsy categorized based on pharmacological and non-pharmacological treatment as 'yes' and 'no' since study diagnosis are reported in this outcome measure. Percentages are rounded-off to the nearest decimal point.
Time Frame: From narcolepsy diagnosis up to study visit (up to 12 months)
Population: SAF contained all enrolled participants who received at least one dose of narcolepsy treatments.
Measure: Number; unit: percentage of participants
Arm/Group | Narcolepsy Type 1 | Narcolepsy Type 2
Number analyzed (Participants) | 157 | 53
percentage of participants
  Pharmacological: No | 5.10 | 7.55
  Pharmacological: Yes | 94.90 | 92.45
  Non-pharmacological: No | 6.37 | 1.89
  Non-pharmacological: Yes | 93.63 | 98.11
Statistical Analysis 1: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Pharmacological; Test type: Superiority; p = 0.5061, Chi-squared
Statistical Analysis 2: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Non-pharmacological; Test type: Superiority; p = 0.2053, Chi-squared

2. Primary Outcome: Percentage of Participants Categorized Based on Non-Pharmacological Treatments Patterns by Treatment Status
Description: Percentage of participants with narcolepsy categorized based on non-pharmacological treatment patterns as 'yes' and 'no' by treatment status [Naïve (untreated) and treated] are reported in this outcome measure. Percentages are rounded-off to the nearest decimal point. Data is collected and reported per Naïve (untreated) and treated arms for this outcome measure.
Time Frame: From narcolepsy diagnosis up to study visit (up to 12 months)
Population: SAF contained all enrolled participants who received at least one dose of narcolepsy treatments.
Measure: Number; unit: percentage of participants
Groups:
- Naive (Untreated): Participants with narcolepsy who were not treated with any pharmacological treatment from diagnosis to study visit (up to 12 months).
- Treated: Participants with narcolepsy who were treated with any pharmacological treatment from diagnosis prior to study visit (up to 12 months).
Arm/Group | Naive (Untreated) | Treated
Number analyzed (Participants) | 12 | 198
percentage of participants
  No | 0 | 5.56
  Yes | 100 | 94.44
Statistical Analysis 1: Comparison: Naive (Untreated) vs Treated; Test type: Superiority; p = 0.4016, Chi-squared

3. Primary Outcome: Percentage of Treated or Naïve (Untreated) Participants for the Type of Pharmacological Treatment Status Since Diagnosis
Description: Percentage of Treated or naïve (Untreated) participants with narcolepsy categorized based on pharmacological treatment status since diagnosis are reported in this outcome measure. Percentages are rounded-off to the nearest decimal point.
Time Frame: From narcolepsy diagnosis up to study visit (up to 12 months)
Population: SAF contained all enrolled participants who received at least one dose of narcolepsy treatments.
Measure: Number; unit: percentage of participants
Arm/Group | Narcolepsy Type 1 | Narcolepsy Type 2
Number analyzed (Participants) | 157 | 53
percentage of participants
  Naive (Untreated) | 5.10 | 7.55
  Treated | 94.90 | 92.45

4. Primary Outcome: Percentage of Participants With the Use of Each Type of Treatment Stratified by Type of Hospital (Public or Private Centers)
Description: Percentages are rounded off to the nearest decimal point.
Time Frame: From a year before narcolepsy diagnosis up to study visit (up to 20 months)
Population: SAF contained all enrolled participants who received at least one dose of narcolepsy treatments. Overall number of participants analyzed is the number of participants available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Narcolepsy Type 1 | Narcolepsy Type 2
Number analyzed (Participants) | 149 | 49
percentage of participants
  Public: Stimulants | 30.60 | 18.92
  Public: Wakefulness-Promoting Agents | 63.43 | 91.89
  Public: Sodium Oxybate | 63.43 | 5.41
  Public: Antidepressants | 34.33 | 5.41
  Public: Benzodiazepines | 8.96 | 0
  Public: Other psychotropic agents | 4.48 | 5.41
  Public: Modafinil + Pitolisant + Sodium Oxybate | 6.72 | 0
  Public: Modafinil + Sodium Oxybate | 16.42 | 0
  Private: Stimulants | 26.67 | 25.00
  Private: Wakefulness-Promoting Agents | 60.00 | 91.67
  Private: Sodium Oxybate | 53.33 | 8.33
  Private: Antidepressants | 26.67 | 33.33
  Private: Benzodiazepines | 0 | 0
  Private: Other psychotropic agents | 0 | 0
  Private: Modafinil + Pitolisant + Sodium Oxybate | 0 | 0
  Private: Modafinil + Sodium Oxybate | 20.00 | 0

5. Secondary Outcome: Number of Participants Categorized by Sociodemographic and Clinical Variables at Study Visit
Description: Sociodemographic variables categorized by age, gender (male/female), ethnicity, educational level ongoing or completed level of education (without studies, primary studies, secondary studies, university studies, other superior studies, not available); occupational status and occupation (student, employed, self-employed, employed but on sick leave due to the study disease, permanent incapacity to work due to the study disease, permanent incapacity to work due to other reasons, unemployed, retired, domestic work, other); civil status (married/with partner, divorced/separated, unmarried, widow/er, unknown); living conditions (alone, wife/husband and/or sons, family caregivers, other caregivers, unknown). Clinical variables categorized by smoking status, alcohol intake, exercise status and family history of narcolepsy in first-degree and second-degree relatives].
Time Frame: Day 1
Population: SAF contained all enrolled participants who received at least one dose of narcolepsy treatments.
Measure: Count of Participants; unit: Participants
Arm/Group | Narcolepsy Type 1 | Narcolepsy Type 2
Number analyzed (Participants) | 157 | 53
Participants
  Age | 157 | 53
  Gender: Male | 78 | 31
  Gender: Female | 79 | 22
  Ethnicity: Caucasian | 147 | 50
  Ethnicity: Hispanic | 7 | 3
  Ethnicity: Asian / Oriental | 1 | 0
  Ethnicity: Other | 2 | 0
  Educational level ongoing or completed level of education: Without studies | 5 | 1
  Educational level ongoing or completed level of education: Primary Studies | 18 | 2
  Educational level ongoing or completed level of education: Secondary Studies | 63 | 21
  Educational level ongoing or completed level of education: University Studies | 56 | 21
  Educational level ongoing or completed level of education: Other Superior Studies | 11 | 5
  Educational level ongoing or completed level of education: Not available | 3 | 3
  Educational level ongoing or completed level of education: Missing | 1 | 0
  Occupational status and occupation: Student | 18 | 2
  Occupational status and occupation: Employed | 82 | 30
  Occupational status and occupation: Self-employed | 12 | 8
  Occupational status and occupation: Employed but on sick leave due to the study disease | 4 | 1
  Occupational status and occupation: Permanent incapacity to work due to the study disease | 10 | 2
  Occupational status and occupation: Permanent incapacity to work due to other reasons | 3 | 1
  Occupational status and occupation: Unemployed | 13 | 4
  Occupational status and occupation: Retired | 9 | 4
  Occupational status and occupation: Domestic work | 3 | 1
  Occupational status and occupation: Other | 2 | 0
  Occupational status and occupation: Missing | 1 | 0
  Civil status: Married/with partner | 72 | 29
  Civil status: Divorced/separated | 12 | 5
  Civil status: Unmarried | 65 | 15
  Civil status: Widow/er | 1 | 1
  Civil status: Unknown | 5 | 3
  Civil status: Missing | 2 | 0
  Living conditions: Alone | 32 | 12
  Living conditions: Wife/Husband and/or sons | 82 | 34
  Living conditions: Family Caregivers | 26 | 1
  Living conditions: Other Caregivers | 2 | 0
  Living conditions: Unknown | 12 | 5
  Living conditions: Missing | 3 | 1
  Smoking status: Current Smoker | 51 | 12
  Smoking status: Ex-Smoker | 33 | 12
  Smoking status: Non-Smoker | 68 | 28
  Smoking status: Unknown | 3 | 1
  Smoking status: Not available | 2 | 0
  Alcohol intake: Never | 75 | 22
  Alcohol intake: Once or less per month | 34 | 12
  Alcohol intake: 2-4 times per month | 25 | 3
  Alcohol intake: 2-3 times per week | 14 | 9
  Alcohol intake: 4 or more times per week | 5 | 4
  Alcohol intake: Unknown | 2 | 1
  Alcohol intake: Not available | 1 | 2
  Alcohol intake: Missing | 1 | 0
  Exercise status: Never | 64 | 16
  Exercise status: Regular | 41 | 25
  Exercise status: Frequently | 29 | 10
  Exercise status: Always | 10 | 0
  Exercise status: Unknown | 8 | 1
  Exercise status: Not available | 5 | 1
  Family history: First-degree relatives | 4 | 4
  Family history: Second-degree relatives | 5 | 1
Statistical Analysis 1: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Educational level ongoing or completed level of education; Test type: Superiority; p = 0.5274, Chi-squared
Statistical Analysis 2: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Occupational status and occupation; Test type: Superiority; p = 0.7051, Chi-squared
Statistical Analysis 3: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Civil status; Test type: Superiority; p = 0.3543, Chi-squared
Statistical Analysis 4: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Living conditions; Test type: Superiority; p = 0.0368, Chi-squared
Statistical Analysis 5: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Smoking status; Test type: Superiority; p = 0.3512, Chi-squared
Statistical Analysis 6: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Alcohol intake; Test type: Superiority; p = 0.1040, Chi-squared
Statistical Analysis 7: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Exercise status; Test type: Superiority; p = 0.0202, Chi-squared
Statistical Analysis 8: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Family history of narcolepsy; Test type: Superiority; p = 0.3503, Chi-squared

6. Secondary Outcome: Height of Participants at Study Visit
Time Frame: Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | Narcolepsy Type 1 | Narcolepsy Type 2
Number analyzed (Participants) | 138 | 50
centimeters (cm) | 168.6 (9.8) | 171.0 (8.7)

7. Secondary Outcome: Weight of Participants at Study Visit
Time Frame: Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Narcolepsy Type 1 | Narcolepsy Type 2
Number analyzed (Participants) | 137 | 50
kilograms (kg) | 77.45 (17.97) | 77.17 (15.08)

8. Secondary Outcome: Body Mass Index (BMI) of Participants at Study Visit
Description: BMI = weight(kg)/height(m)^2
Time Frame: Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: kilograms per meters square (kg/m^2)
Arm/Group | Narcolepsy Type 1 | Narcolepsy Type 2
Number analyzed (Participants) | 137 | 50
kilograms per meters square (kg/m^2) | 27.18 (5.58) | 26.34 (4.71)

9. Secondary Outcome: Blood Pressure (BP) of Participants at Study Visit
Time Frame: Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mm Hg)
Arm/Group | Narcolepsy Type 1 | Narcolepsy Type 2
Number analyzed (Participants) | 72 | 28
millimeters of mercury (mm Hg)
  Systolic BP | 121.0 (16.4) | 120.0 (14.1)
  Diastolic BP | 75.7 (12.8) | 74.3 (10.9)

10. Secondary Outcome: Percentage of Participants Categorized Based on Different Specialists Who Diagnosed Narcolepsy
Description: Specialist who diagnosed narcolepsy were categorized as general practitioners, neurologist, neuropediatrician, neurophysiologist, pneumologist, somnologist, somnologist-unit and specialist (Not specified). Percentage of participants are rounded-off to the nearest decimal point.
Time Frame: From a year before narcolepsy diagnosis up to study visit (up to 20 months)
Population: SAF contained all enrolled participants who received at least one dose of narcolepsy treatments. Overall number of participants analyzed is the number of participants available for analysis. Number analyzed is the number of participants with data available for the specified categories.
Measure: Number; unit: percentage of participants
Arm/Group | Narcolepsy Type 1 | Narcolepsy Type 2
Number analyzed (Participants) | 156 | 53
percentage of participants
  General practitioner | 1.28 | 5.66
  Neurologist | 37.18 | 24.53
  Neuropediatrician | 1.92 | 0
  Neurophysiologist | 49.36 | 43.40
  Pneumologist | 2.56 | 18.87
  Somnologist | 3.21 | 7.55
  Somnologist-unit | 3.85 | 0
  Specialist (Not specified) | 0.64 | 0
Statistical Analysis 1: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; General practitioner; Test type: Superiority; p = 0.0715, Chi-squared
Statistical Analysis 2: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Neurologist; Test type: Superiority; p = 0.0929, Chi-squared
Statistical Analysis 3: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Neuropediatrician; Test type: Superiority; p = 0.3092, Chi-squared
Statistical Analysis 4: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Neurophysiologist; Test type: Superiority; p = 0.4528, Chi-squared
Statistical Analysis 5: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Pneumologist; Test type: Superiority; p < 0.0001, Chi-squared
Statistical Analysis 6: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Somnologist; Test type: Superiority; p = 0.1785, Chi-squared
Statistical Analysis 7: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Somnologist-unit; Test type: Superiority; p = 0.1474, Chi-squared

11. Secondary Outcome: Percentage of Participants Categorized Based on Usage of Different Procedures or Tests for the Diagnosis of Narcolepsy
Description: Different procedures or tests for diagnosis included clinical history, Clinical Assessment: Epworth sleepiness scale (ESS) [ESS consists of 8 items, on a 4-point scale (0-3) ranging from "0=No chance of dozing" to "3=High chance of dozing" while engaged in eight different activities. The score can range from 0 to 24. Higher scores indicate stronger subjective daytime sleepiness, and scores below 10 are within the normal range], Neurological Assessment, Multiple sleep latency test (MSLT), Apnea-hypopnea index (AHI), Other procedures, Human leucocyte antigen (HLA) typing, Hypocretin-1 cerebrospinal fluid (CSF) or Orexin. Percentages are rounded-off to the nearest decimal point.
Time Frame: From a year before narcolepsy diagnosis up to 12 months
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Narcolepsy Type 1 | Narcolepsy Type 2
Number analyzed (Participants) | 143 | 45
percentage of participants
  Clinical History | 91.08 | 84.91
  Clinical Assessment: Epworth sleepiness scale (ESS) | 54.14 | 58.49
  Neurological Assessment | 59.87 | 43.40
  Multiple sleep latency test (MSLT) | 96.18 | 90.57
  Apnea-hypopnea index (AHI) | 52.87 | 45.28
  Other procedures | 7.64 | 9.43
  Human leucocyte antigen (HLA) typing | 51.59 | 32.08
  Hypocretin-1 cerebrospinal fluid (CSF) or Orexin | 6.37 | 0
Statistical Analysis 1: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Clinical history; Test type: Superiority; p = 0.2042, Chi-squared
Statistical Analysis 2: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Clinical assessment: ESS; Test type: Superiority; p = 0.5818, Chi-squared
Statistical Analysis 3: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Neurological assessment; Test type: Superiority; p = 0.0368, Chi-squared
Statistical Analysis 4: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; MSLT; Test type: Superiority; p = 0.1128, Chi-squared
Statistical Analysis 5: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; AHI; Test type: Superiority; p = 0.3396, Chi-squared
Statistical Analysis 6: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Other procedures; Test type: Superiority; p = 0.6794, Chi-squared
Statistical Analysis 7: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; HLA typing; Test type: Superiority; p = 0.0138, Chi-squared
Statistical Analysis 8: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Hypocretin-1 CSF or Orexin; Test type: Superiority; p = 0.0597, Chi-squared

12. Secondary Outcome: Time From First Symptom to Diagnosis of Narcolepsy
Description: Time from first symptom in participant to diagnosis is the time when the first symptom of narcolepsy was identified until its diagnosis during retrospective visit. As the first symptom and the diagnosis at retrospective visit could be any time in the past up to end of enrolment in this study. Thus, as pre-planned data for this outcome measure may exceed the duration of the study.
Time Frame: From first symptom of narcolepsy up to diagnosis maximum up to 59.92 years (retrospective data was retrieved and observed during 20 months of this study)
Population: as for outcome 4
Measure: Median (Full Range); unit: years
Arm/Group | Narcolepsy Type 1 | Narcolepsy Type 2
Number analyzed (Participants) | 139 | 40
years | 6.30 [0.00 to 59.92] | 2.94 [0.00 to 47.87]
Statistical Analysis 1: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Test type: Superiority; p = 0.1171, t-test, 2 sided

13. Secondary Outcome: Time From Diagnosis of Narcolepsy to First Treatment
Description: Time from diagnosis to first treatment is the time required to diagnose the first symptom of narcolepsy until the first treatment is provided after diagnosis retrospectively. As the first symptom and the diagnosis at retrospective visit could be any time in the past up to end of enrolment in this study. Thus, as pre-planned data for this outcome measure may exceed the duration of the study.
Time Frame: From first symptom of narcolepsy up to diagnosis maximum up to 46.04 years (retrospective data was retrieved and observed during 20 months of this study)
Population: as for outcome 4
Measure: Median (Full Range); unit: years
Arm/Group | Narcolepsy Type 1 | Narcolepsy Type 2
Number analyzed (Participants) | 152 | 49
years | 0.05 [0.00 to 46.04] | 0.02 [0.00 to 4.43]
Statistical Analysis 1: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Test type: Superiority; p = 0.3834, t-test, 2 sided

14. Secondary Outcome: Percentage of Participants Categorized Based on Pharmacological Treatment and Interventions Received in Relation With the Presence of Most Typical Symptoms
Time Frame: From a year before narcolepsy diagnosis up to study visit (up to 20 months)
Population: Analysis population included all eligible participants whose data was retrieved and analyzed. Data was not collected for this outcome measure as data was not available in the medical records.
Arm/Group | Narcolepsy Type 1 | Narcolepsy Type 2
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Percentage of Participants With Pharmacological Treatments at Each Line
Description: Pharmacological Treatments were categorized as 1st treatment after diagnosis (monotherapy and combinations), treatments used from diagnosis to study visit and treatments at study visit (monotherapy and combinations). Percentages are rounded off to the nearest decimal point.
Time Frame: From a year before narcolepsy diagnosis up to study visit (up to 20 months)
Population: SAF contained all enrolled participants who received at least one dose of narcolepsy treatments.
Measure: Number; unit: percentage of participants
Arm/Group | Narcolepsy Type 1 | Narcolepsy Type 2
Number analyzed (Participants) | 157 | 53
percentage of participants
  1st Treatment: Monotherapy | 82.80 | 90.57
  1st Treatment: Combinations | 12.10 | 1.89
  From Diagnosis up to Study Visit | 94.90 | 92.45
  At Study Visit: Monotherapy | 54.14 | 71.70
  At Study Visit: Combinations | 24.94 | 11.32

16. Secondary Outcome: Sustained Attention to Response Task (SART)
Description: Behavioral measure of working memory, attention, and impulse/inhibitory control - The Sustained Attention to Response Task (SART) is a computer-based go/no-go task that requires participants to withhold behavioral response to a single, infrequent target (often the digit 3) presented amongst a background of frequent non-targets (0-2, 4-9). After each block, two probe questions are presented in succession. The first asks, "Where was your attention focused during this block of trials?" Participants respond on a 6-point Likert scale, where 1 represents, "on task," and 6, "off task." A second question asks, "How aware were you of where your attention was during this block of trials?" Participants respond on a similar scale, where 1 represents, "aware," and 6, "unaware."
Time Frame: From a year before narcolepsy diagnosis up to study visit (up to 20 months)
Population: as for outcome 14
Arm/Group | Narcolepsy Type 1 | Narcolepsy Type 2
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Maintenance of Wakefulness Test (MWT)
Description: The MWT is a validated objective measure that evaluates a person's ability to remain awake under soporific conditions for a defined period of time. This tendency to fall asleep is measured via electroencephalography-derived sleep latency. Sleep onset is defined as the first epoch of greater than 15 seconds of cumulative sleep in a 30-second epoch. During each MWT session (1 session = 40 minutes), participants will be instructed to sit quietly and remain awake for as long as possible. If no sleep has been observed according to these rules, then the latency is defined as 40 minutes. MWT sleep latency ranges from 0 to 40 minutes, with higher scores indicating greater ability to stay awake.
Time Frame: From a year before narcolepsy diagnosis up to study visit (up to 20 months)
Population: as for outcome 14
Arm/Group | Narcolepsy Type 1 | Narcolepsy Type 2
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Epworth Sleepiness Scale (ESS)
Description: ESS is a subjective, self-administered questionnaire to assess daytime sleepiness and consists of 8 items, on a 4-point scale (0-3) ranging from "No chance of dozing" to "High chance of dozing" while engaged in eight different activities. The score can range from 0 to 24. Higher scores indicate stronger subjective daytime sleepiness, and scores below 10 are considered to be within the normal range.
Time Frame: From a year before narcolepsy diagnosis up to 12 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Narcolepsy Type 1 | Narcolepsy Type 2
Number analyzed (Participants) | 75 | 31
score on a scale | 18.08 (3.51) | 16.35 (4.29)
Statistical Analysis 1: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Test type: Superiority; p = 0.0531, t-test, 2 sided

19. Secondary Outcome: Percentage of Participants Categorized Based on Different Non-pharmacological Treatment Approach
Description: Non-pharmacological treatment approach was categorized as take short naps, maintain a regular sleep schedule, avoid caffeine or alcohol before bedtime, avoid smoking, especially at night, exercise daily, avoid large, heavy meals right before bedtime, and other. Percentage of participants are rounded-off to the nearest decimal point.
Time Frame: From a year before narcolepsy diagnosis up to study visit (up to 20 months)
Population: SAF contained all enrolled participants who received at least one dose of narcolepsy treatments.
Measure: Number; unit: percentage of participants
Arm/Group | Narcolepsy Type 1 | Narcolepsy Type 2
Number analyzed (Participants) | 157 | 53
percentage of participants
  Take short naps | 79.62 | 60.38
  Maintain a regular sleep schedule | 68.15 | 69.81
  Avoid caffeine or alcohol before bedtime | 56.69 | 47.17
  Avoid smoking, especially at night | 36.94 | 37.74
  Exercise daily | 36.31 | 30.19
  Avoid large, heavy meals right before bedtime | 57.96 | 62.26
  Other | 10.19 | 13.21
Statistical Analysis 1: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Take short naps; Test type: Superiority; p = 0.0005, Chi-squared
Statistical Analysis 2: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Maintain a regular sleep schedule; Test type: Superiority; p = 0.8221, Chi-squared
Statistical Analysis 3: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Avoid caffeine or alcohol before bedtime; Test type: Superiority; p = 0.2291, Chi-squared
Statistical Analysis 4: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Avoid smoking, especially at night; Test type: Superiority; p = 0.9177, Chi-squared
Statistical Analysis 5: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Exercise daily; Test type: Superiority; p = 0.4188, Chi-squared
Statistical Analysis 6: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Avoid large, heavy meals right before bedtime; Test type: Superiority; p = 0.5818, Chi-squared
Statistical Analysis 7: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Other; Test type: Superiority; p = 0.5432, Chi-squared

20. Secondary Outcome: Percentage of Participants Categorized Based on Utilization of Direct Healthcare Resource Utilized Per Year
Description: Direct healthcare resource utilized per year were categorized as treatments for narcolepsy, routine monitoring visits, tests, emergency visits, hospitalizations and complications associated to narcolepsy. Percentage of participants are rounded-off to the nearest decimal point.
Time Frame: From a year before study visit (up to 12 months)
Population: SAF contained all enrolled participants who received at least one dose of narcolepsy treatments.
Measure: Number; unit: percentage of participants
Arm/Group | Narcolepsy Type 1 | Narcolepsy Type 2
Number analyzed (Participants) | 157 | 53
percentage of participants
  Treatment | 89.81 | 86.79
  Routine monitoring visits | 78.34 | 64.15
  Clinical Tests | 78.98 | 64.15
  Emergency visits | 1.27 | 1.89
  Hospitalizations | 0 | 1.89
  Complications | 9.55 | 5.66
Statistical Analysis 1: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Treatment; Test type: Superiority; p = 0.5432, Chi-squared
Statistical Analysis 2: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Routine monitoring visits; Test type: Superiority; p = 0.0397, Chi-squared
Statistical Analysis 3: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Tests; Test type: Superiority; p = 0.0306, Chi-squared
Statistical Analysis 4: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Emergency visits; Test type: Superiority; p = 0.7451, Chi-squared
Statistical Analysis 5: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Hospitalizations; Test type: Superiority; p = 0.0845, Chi-squared
Statistical Analysis 6: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Complications; Test type: Superiority; p = 0.3813, Chi-squared

21. Secondary Outcome: Duration of Hospitalization
Description: Duration of hospitalization is the total number of days at which participants were admitted in hospital.
Time Frame: From a year before study visit (up to 12 months)
Population: SAF contained all enrolled participants who received at least one dose of narcolepsy treatments. Overall number of participants analyzed is the number of participants who were hospitalized.
Measure: Median (Full Range); unit: days
Arm/Group | Narcolepsy Type 1 | Narcolepsy Type 2
Number analyzed (Participants) | 0 | 1
days |  | 1.00 [1 to 1]

22. Secondary Outcome: Work Productivity and Activity Impairment (WPAI) Score
Description: The WPAI is a questionnaire that assesses the impact of an intervention on work productivity, evaluating 4 areas including absenteeism [Q2/(Q2+Q4)], presenteeism [Q5/10], work productivity loss {Q2/(Q2+Q4)+[(1-(Q2/(Q2+Q4))x(Q5/10)]}, and activity impairment [Q6/10], calculated based on three items: (Q2) the number of hours missed from work due to health problems in the past seven days; (Q4) the number of actual work hours in the past seven days; and (Q5) to what degree did the disease impair the productivity while working past seven days. The data calculated for each area is then converted to percent. Each of the areas is scored separately as a percentage, ranging from 0 to 100, with higher scores indicating greater impairment and less productivity.
Time Frame: From a year before study visit (up to 20 months)
Population: SAF contained all enrolled participants who received at least one dose of narcolepsy treatments. Overall number of participants analyzed is the number of participants available for analysis. Number analyzed is the number of participants available for analysis in the specified categories.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Narcolepsy Type 1 | Narcolepsy Type 2
Number analyzed (Participants) | 91 | 36
score on a scale
  Absenteeism: number analyzed (Participants) | 89 | 36
  Absenteeism | 11.57 (25.24) | 3.23 (8.87)
  Presenteeism: number analyzed (Participants) | 85 | 36
  Presenteeism | 32.4 (29.5) | 28.1 (29.8)
  Work Productivity Loss: number analyzed (Participants) | 85 | 36
  Work Productivity Loss | 34.63 (30.97) | 29.54 (30.73)
  Activity Impairment / Disability | 36.2 (31.4) | 31.1 (31.8)
Statistical Analysis 1: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Absenteeism; Test type: Superiority; p = 0.0034, t-test, 2 sided
Statistical Analysis 2: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Presenteeism; Test type: Superiority; p = 0.2178, t-test, 2 sided
Statistical Analysis 3: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Work productivity loss; Test type: Superiority; p = 0.1758, t-test, 2 sided
Statistical Analysis 4: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Activity Impairment / disability; Test type: Superiority; p = 0.1789, t-test, 2 sided

23. Secondary Outcome: Number of Participants Categorized Based on Occupational Accidents
Time Frame: From a year before study visit (up to 20 months)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Narcolepsy Type 1 | Narcolepsy Type 2
Number analyzed (Participants) | 139 | 53
Participants
  No | 131 | 51
  Yes | 8 | 2
Statistical Analysis 1: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Test type: Superiority; p = 0.5806, Chi-squared

24. Secondary Outcome: Percentage of Participants Categorized Based on Cost of Direct Healthcare Resources Utilized by Participants Per Year
Description: Cost of direct healthcare resources utilized by participants per year based on costs of following direct healthcare resources was to be included: treatment received, routine monitoring visits (specialists and GPs), tests performed, emergency rooms visits, hospitalizations and complications derived from narcolepsy, and unitary costs.
Time Frame: From a year before study visit (approximately 20 months)
Population: as for outcome 14
Arm/Group | Narcolepsy Type 1 | Narcolepsy Type 2
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: Percentage of Participants With Health Related Quality of Life (HRQoL) Assessed by European Quality of Life Five Dimension (EQ-5D) Questionnaire
Description: The EQ-5D questionnaire is a generic instrument for describing and valuing health. It is based on a descriptive system that defines health in terms of 5 dimensions: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Each dimension has 3 response categories corresponding to no problems, some problems, and extreme problems. The instrument is designed for self-completion, and respondents also rate their overall health on the day of the interview on a 0-100 hash-marked, vertical visual analogue scale (EQ-VAS). Higher score indicates better health state. Percentage of participants are rounded-off to the nearest decimal point.
Time Frame: From a year before narcolepsy diagnosis up to study visit (up to 20 months)
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Narcolepsy Type 1 | Narcolepsy Type 2
Number analyzed (Participants) | 149 | 53
percentage of participants
  Mobility: I have no problems in walking about | 85.91 | 84.91
  Mobility: I have slight problems in walking about | 8.05 | 15.09
  Mobility: I have moderate problems in walking about | 4.70 | 0
  Mobility: I have severe problems in walking about | 1.34 | 0
  Mobility: I am unable to walk about | 0 | 0
  Self-Care: I have no problems washing or dressing myself | 93.96 | 90.57
  Self-Care: I have slight problems washing or dressing myself | 4.69 | 9.43
  Self-Care: I have moderate problems washing or dressing myself | 0.70 | 0
  Self-Care: I have severe problems washing or dressing myself | 0.70 | 0
  Self-Care: I am unable to wash or dress myself | 0 | 0
  Usual activities: I have no problems doing my usual activities | 51.01 | 58.49
  Usual activities: I have slight problems doing my usual activities | 17.45 | 24.53
  Usual activities: I have moderate problems doing my usual activities | 24.83 | 16.98
  Usual activities: I have severe problems doing my usual activities | 6.71 | 0
  Usual activities: I am unable to do my usual activities | 0 | 0
  Pain / Discomfort: I have no pain or discomfort | 63.09 | 67.92
  Pain / Discomfort: I have slight pain or discomfort | 17.45 | 13.21
  Pain / Discomfort: I have moderate pain or discomfort | 12.08 | 16.98
  Pain / Discomfort: I have severe pain or discomfort | 7.38 | 1.89
  Pain / Discomfort: I have extreme pain or discomfort | 0 | 0
  Anxiety / Depression: I am not anxious or depressed | 48.99 | 52.83
  Anxiety / Depression: I am slightly anxious or depressed | 26.18 | 20.75
  Anxiety / Depression: I am moderately anxious or depressed | 18.79 | 20.75
  Anxiety / Depression: I am severely anxious or depressed | 4.03 | 5.66
  Anxiety / Depression: I am extremely anxious or depressed | 2.01 | 0
Statistical Analysis 1: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Mobility; Test type: Superiority; p = 0.1602, Chi-squared
Statistical Analysis 2: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Self-Care; Test type: Superiority; p = 0.5249, Chi-squared
Statistical Analysis 3: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Usual activities; Test type: Superiority; p = 0.1095, Chi-squared
Statistical Analysis 4: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Pain / Discomfort; Test type: Superiority; p = 0.3528, Chi-squared
Statistical Analysis 5: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Anxiety / Depression; Test type: Superiority; p = 0.7434, Chi-squared

26. Secondary Outcome: Stigma Scale for Chronic Illness 8-item Version (SSCI-8) Total Score
Description: SSCl-8 is an 8 items scale (2 items measuring internalized stigma, 5 items measuring enacted stigma, and 1 item, which exhibited split loading, measuring either or both internalized and enacted stigma) developed to assess internalized and enacted/experienced stigma across neurological conditions. It uses a 5-point Likert scale ranging from 1 (never) to 5 (always) for scoring each item. The total score is calculated by summing individual items, ranging from 8 to 40. Higher scores indicate worsening of condition.
Time Frame: From a year before narcolepsy diagnosis up to study visit (up to 20 months)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Narcolepsy Type 1 | Narcolepsy Type 2
Number analyzed (Participants) | 149 | 58
score on a scale | 15.5 (6.1) | 14.1 (5.5)
Statistical Analysis 1: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Test type: Superiority; p = 0.0396, t-test, 2 sided

27. Secondary Outcome: Treatment Satisfaction of Participants Assessed by Treatment Satisfaction Questionnaire for Medication (TSQM-9)
Description: TSQM-9 measures participant satisfaction with the medication in 3 domains: Effectiveness, convenience, and global satisfaction. The scores were computed by adding items for each domain, i.e., 1 to 3 for effectiveness, 4 to 6 for convenience, and 7 to 9 for global satisfaction. The lowest possible score (1 for each item and 3 for all 3 subscales) was subtracted from the composite score and divided by the greatest possible score range. The greatest range was (7-1) x 3 items = 18 for effectiveness and convenience, and (5-1) x 3 items = 12 for global satisfaction. This provided a transformed score between 0 and 1 that was then multiplied by 100. TSQM-9 domain scores range from 0 to 100, with higher scores indicating greater satisfaction for that domain.
Time Frame: From a year before narcolepsy diagnosis up to study visit (up to 20 months)
Population: SAF contained all enrolled participants who received at least one dose of narcolepsy treatments. Overall number of participants analyzed is the number of participants available for analysis. Number analyzed is the number of participants available for analysis in the specified data set.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Narcolepsy Type 1 | Narcolepsy Type 2
Number analyzed (Participants) | 141 | 46
score on a scale
  Effectiveness | 67.53 (19.12) | 63.05 (21.19)
  Convenience: number analyzed (Participants) | 140 | 46
  Convenience | 74.21 (19.99) | 73.06 (16.41)
  Global Satisfaction | 68.54 (20.33) | 63.36 (24.92)
Statistical Analysis 1: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Effectiveness; Test type: Superiority; p = 0.0394, t-test, 2 sided
Statistical Analysis 2: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Convenience; Test type: Superiority; p = 0.3093, t-test, 2 sided
Statistical Analysis 3: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Global satisfaction; Test type: Superiority; p = 0.2296, t-test, 2 sided

28. Secondary Outcome: Percentages of Participants Based on Most Prevalent Comorbidities and Other Concomitant Disorders Associated With Narcolepsy
Description: Percentage of participants are rounded-off to the nearest decimal point.
Time Frame: From a year before narcolepsy diagnosis up to study visit (up to 20 months)
Population: SAF contained all enrolled participants who received at least one dose of narcolepsy treatments.
Measure: Number; unit: percentage of participants
Arm/Group | Narcolepsy Type 1 | Narcolepsy Type 2
Number analyzed (Participants) | 157 | 53
percentage of participants
  Depression | 14.65 | 7.55
  Bipolar disorder | 0 | 1.89
  Anxiety disorders | 12.74 | 7.55
  Post-traumatic stress disorder | 0 | 0
  Panic disorder | 0 | 1.89
  Phobia disorder | 0.64 | 0
  Obsessive compulsive disorder | 0.64 | 0
  Diagnosis of attention deficit hyperactivity disorder (ADHD) | 1.91 | 0
  Obesity | 22.29 | 15.09
  Endocrine disorders | 7.01 | 9.43
  Myocardial Infarction | 0 | 0
  Urinary Incontinence | 0 | 0
  Congestive heart failure (CHF) | 0 | 0
  Peripheral vascular disease | 1.27 | 0
  Cardiovascular accident or transient ischemic attack (TIA) | 0.64 | 0
  Dementia | 0 | 0
  Chronic obstructive pulmonary disease (COPD) | 0.64 | 0
  Connective tissue disease | 0.64 | 0
  Peptic ulcer disease | 0 | 0
  Liver Disease | 1.27 | 1.89
  Diabetes Mellitus | 1.91 | 0
  Hemiplegia | 0 | 0
  Moderate to severe chronic kidney disease (CKD) | 0 | 0
  Solid tumor | 2.55 | 0
  Leukemia | 0 | 0
  Lymphoma | 0 | 0
  Acquired Immunodeficiency Syndrome (AIDS) | 0.64 | 0
  Others | 17.20 | 9.43
Statistical Analysis 1: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Depression; Test type: Superiority; p = 0.1817, Chi-squared
Statistical Analysis 2: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Bipolar disorder; Test type: Superiority; p = 0.0885, Chi-squared
Statistical Analysis 3: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Anxiety disorders; Test type: Superiority; p = 0.3043, Chi-squared
Statistical Analysis 4: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Panic disorder; Test type: Superiority; p = 0.0885, Chi-squared
Statistical Analysis 5: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Phobia disorder; Test type: Superiority; p = 0.5603, Chi-squared
Statistical Analysis 6: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Obsessive compulsive disorder; Test type: Superiority; p = 0.5603, Chi-squared
Statistical Analysis 7: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Diagnosis of ADHD; Test type: Superiority; p = 0.3646, Chi-squared
Statistical Analysis 8: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Obesity; Test type: Superiority; p = 0.2615, Chi-squared
Statistical Analysis 9: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Endocrine Disorders; Test type: Superiority; p = 0.3076, Chi-squared
Statistical Analysis 10: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Peripheral vascular disease; Test type: Superiority; p = 0.4090, Chi-squared
Statistical Analysis 11: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Cardiovascular accident or transient ischemic attack (TIA); Test type: Superiority; p = 0.5603, Chi-squared
Statistical Analysis 12: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; COPD; Test type: Superiority; p = 0.5603, Chi-squared
Statistical Analysis 13: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Connective tissue disease; Test type: Superiority; p = 0.5603, Chi-squared
Statistical Analysis 14: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Liver Disease; Test type: Superiority; p = 0.7451, Chi-squared
Statistical Analysis 15: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Diabetes Mellitus; Test type: Superiority; p = 0.3108, Chi-squared
Statistical Analysis 16: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Solid Tumor; Test type: Superiority; p = 0.2407, Chi-squared
Statistical Analysis 17: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; AIDS; Test type: Superiority; p = 0.5603, Chi-squared
Statistical Analysis 18: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Others; Test type: Superiority; p = 0.1739, Chi-squared

29. Secondary Outcome: Charlson Comorbidity Index (CCI)
Description: CCI is a scale to estimate 10-year mortality based on a score from a range of 12 comorbidities, the comorbidity score ranges from 0 to a maximum of 24 points. Higher scores indicate the higher chances of mortality.
Time Frame: From a year before narcolepsy diagnosis up to study visit (up to 20 months)
Population: SAF contained all enrolled participants who received at least one dose of narcolepsy treatments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Narcolepsy Type 1 | Narcolepsy Type 2
Number analyzed (Participants) | 157 | 53
score on a scale | 0.4 (1.1) | 0.2 (0.7)
Statistical Analysis 1: Comparison: Narcolepsy Type 1 vs Narcolepsy Type 2; Test type: Superiority; p = 0.3585, t-test, 2 sided

30. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant administered a medicinal product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, a new disease or worsening in severity or frequency of a concomitant disease, temporally associated with the use of a medicinal product, whether or not the event is considered causally related to the use of the product.
Time Frame: Up to 20 months
Population: SAF contained all enrolled participants who received at least one dose of narcolepsy treatments. As pre-specified in the protocol and statistical analysis plan (SAP) the adverse events were collected for overall participants who received any narcolepsy treatment (Pharmacological or non-pharmacological) irrespective of the narcolepsy type.
Measure: Count of Participants; unit: Participants
Groups:
- Overall: Participants who received any narcolepsy treatment (Pharmacological or non-pharmacological) since diagnosis to study visit (up to 12 months).
Arm/Group | Overall
Number analyzed (Participants) | 210
Participants | 11

ADVERSE EVENTS:
Time Frame: Up to 20 months
Description: SAF contained all enrolled participants who received at least one dose of narcolepsy treatments. As pre-specified in the protocol and SAP the adverse events were collected for overall participants who received any narcolepsy treatment (Pharmacological or non-pharmacological) irrespective of the narcolepsy type.
Arm/Group | Overall
All-Cause Mortality (participants affected / at risk) | 0/210
Serious Adverse Events (participants affected / at risk) | 0/210
Other Adverse Events (participants affected / at risk) | 11/210
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall (N=210)
Tachycardia (Cardiac disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Cell death (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Enuresis (Psychiatric disorders) | 1
Nervousness (Psychiatric disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-09-02): https://cdn.clinicaltrials.gov/large-docs/38/NCT04667338/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-19): https://cdn.clinicaltrials.gov/large-docs/38/NCT04667338/SAP_001.pdf